CLINICAL TRIAL: NCT04715373
Title: Less Invasive Administration of Surfactant in the Delivery Room for Extremely Preterm Infants: A Randomized Control Trial
Brief Title: LISA in the Delivery Room for Extremely Preterm Infants
Acronym: DRLISA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Chiesi USA, Inc. (Industry)
Responsible Party: Principal Investigator, Venkat Kakkilaya, Associate Professor of Pediatrics, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2020-0926
Record Dates: First submitted 2021-01-13; First posted 2021-01-20 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Extreme Prematurity; Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DR-LISA (Experimental): Experimental:
  Group 1: (Intervention Arm) Infants will be resuscitated per NRP guidelines. Infant with stable HR and respiratory effort will be changed to binasal prongs. A trained physician will perform LISA. Infant will be maintained on CPAP by prongs during the procedure. . PPV will be provided if needed after the procedure. Infants requiring FiO2 >0.8 on CPAP 8 cm H2O to maintain SpO2 88-94% by 20 minutes of life will be intubated prior to transport. After admission to the NICU, CPAP will be titrated 5-8 cm H2O.
  Interventions: Procedure: LISA
- NICU-LISA (Active Comparator): Group 2: Control Arm Infants will be resuscitated per NRP guidelines. Infant with stable HR and respiratory effort will be changed to binasal prongs and transported to NICU on CPAP. After admission to NICU, CPAP will be escalated every 30 minutes up to a maximum level of 7 cm H2O at which point infant would qualify for LISA if the FiO2 requirement is ≥0.3. Infants requiring FiO2 >0.8 to maintain SpO2 88-94% by 20 minutes of life will be intubated in the DR.
  Interventions: Procedure: LISA

INTERVENTIONS:
Procedure: LISA — LISA administered in the DR after initial resuscitation or in the NICU after stepwise escalation of CPAP based on FiO2 ≥0.3. While maintaining infant on CPAP with binasal prongs/small nasal mask, a thin catheter (Hobart method) is inserted below the vocal cord using direct laryngoscopy. Poractant alfa (200mg/kg) is administered slowly over 2-3 minutes. Catheter is then withdrawn and infant is maintained on CPAP

SUMMARY:
The purpose of this study is to evaluate the effect of LISA used in the delivery room (DR) in decreasing the intubation rates in preterm infants at 22-25 weeks gestational age (GA), during first 72 hours compared to the standard approach of stabilization on nasal CPAP in the DR and administering surfactant in the NICU.

Infants in both groups will be resuscitated per NRP algorithm. Infants who maintain a stable HR and respiratory effort on CPAP will qualify for the intervention. Infants in Group 1 (Intervention arm) will receive LISA in DR. CPAP will be titrated between 5-8 cm H20 after LISA. Infants in Group 2 (Control arm) will be transferred to NICU on CPAP. The CPAP level will be increased stepwise every 30 minutes to 7 cm H2O if FiO2 ≥0.3. Infants requiring CPAP 7 at FiO2 ≥0.3 will receive LISA. CPAP will be titrated between 5-8 cm H20 after LISA.

Infants in both arms requiring CPAP 7 and FiO2 >0.8 at 20 MOL in the delivery room will be intubated in DR. Any infant with a heart rate not responding with appropriate PPV will be intubated in the DR. CXR will be obtain on admission and umbilical lines will be placed. Infants in both arm who require FiO2 ≥0.6 for ≥1 hour, apnea requiring stimulation 3 times within one hour or ≥6 over 6 hour period, any apnea requiring PPV, or CO2 >0.65 in two consecutive blood gases drawn over two hours will be considered as reasons for intubation after LISA.

Primary outcome is the need for MV within 72 hours of life, secondary outcome includes need for MV during first week of life and during hospital stay, bronchopulmonary dysplasia (BPD), intraventricular hemorrhage (IVH), necrotizing enterocolitis (NEC), spontaneous intestinal perforation (SIP), need for treatment of patent ductus arteriosus (PDA), composite death or BPD and mortality. This is a feasibility trial with the intention to enroll 30 infants in each arm of the study over three years.

DETAILED DESCRIPTION:
This is a single center, unblinded, randomized control, feasibility trial to evaluate the use of LISA in the DR for extremely preterm infants born 22-25 weeks GA who were successfully resuscitated without being intubated. The study team will approach a mother who is at risk of delivering an infant between 22-25 week GA for consent to be included in the study. Infants will be resuscitated according to NRP algorithm. Infants who are successfully resuscitated without requiring intubation and mechanical ventilation (HR >100, regular spontaneous respiratory effort, able to maintain oxygenation per NRP target saturation goal) are eligible for enrollment. Randomization will be achieved by opening an opaque envelope.

* Intervention arm (DR-LISA): Infants with a stable heart rate and spontaneous respiratory effort on CPAP are eligible for surfactant therapy. A LISA catheter will be prepared for use prior to the birth of the infant. Surfactant will be drawn into a syringe soon after the initial stabilization. A trained physician will perform LISA. The infant will be maintained on CPAP by prongs during the procedure. PPV will be provided if needed after the procedure. The infant will be monitored in the DR for stable HR, respiration and SpO2 prior to being moved to a transporter. Infants requiring FiO2 >0.8 on CPAP 8 cm H2O to maintain SpO2 88-94% by 20 minutes of life will be intubated prior to transport. After admission to NICU, CPAP level will be titrated between 5-8 cm H20 based on FiO2 threshold ≥0.3
* Control arm: Infants will be resuscitated per NRP guidelines. Infant with stable HR and respiratory effort will be changed to binasal prongs and transported to NICU on CPAP. CPAP level be titrated between 5- 7 cm H2O in the DR. Infants requiring FiO2 >0.8 to maintain SpO2 88-94% by 20 minutes of life will be intubated in DR. After admission to NICU, CPAP will be escalated every 30 minutes up to a maximum level of 7 cm H2O at which point infant would qualify for LISA if the FiO2 requirement is ≥0.3. CPAP level will be titrated between 5-8 cm H20 based on FiO2 threshold ≥0.3. Infants in both groups who require FiO2 ≥0.6 for ≥1 hour, apnea requiring stimulation 3 times within one hour or ≥6 over 6 hour period, any apnea requiring PPV, or CO2 >0.65 in two consecutive blood gases drawn over two hours will be considered as reasons for intubation after LISA.

Repeat doses of surfactant will be administered every 12 hours for FiO2 ≥0.4 up to a maximum of three doses.

ELIGIBILITY:
Inclusion Criteria:

* Infants born 22 -25 weeks GA
* Resuscitated without requiring intubation and maintaining HR >100, and spontaneous respiratory effort on CPAP 5-7 cm H2O)

Exclusion Criteria:

* Major congenital anomalies
* Infants receiving only comfort care
* Mothers with impaired decision making capacity

Ages: 5 Minutes to 20 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Need for intubation and/any mechanical ventilation | within 72 hours of life
  Any Infant randomized to the study requiring intubation and/mechanical ventilation

SECONDARY OUTCOMES:
Need for mechanical ventilation within 7 days of life | Within 7 days of life.
  Any Infant randomized to the study requiring intubation and/mechanical ventilation
Mechanical Ventilation | Until hospital discharge or 6 months of life
  Any infant requiring MV
High Frequency Ventilation | Until hospital discharge or 6 month of life
  Any infant requiring high frequency ventilation. This outcome will not be analyzed because of a protocol amendment.
Mechanical ventilator days | Until hospital discharge or 6 months of life
  Infant requiring MV for longer than 12 hours in a day
Bronchopulmonary dysplasia | Until hospital discharge or 6 months of life
  Infant requiring supplemental oxygen at 36 weeks PMA
Severe intraventricular hemorrhage | Until hospital discharge or 6 months of life
  Grade 3 or 4 intraventricular hemorrhage
Pneumothorax | Until hospital discharge or 6 months of life
  Radiographic evidence of pneumothorax
Desaturation (SpO2 <80) and Bradycardia (HR <100) events | During the first 72 hours
  Any desaturation and bradycardia event lasting >10 seconds during LISA procedure
Proportion of infants requiring >1 LISA attempt | During the first 72 hours of life
  Any direct laryngoscopy attempt
Death or BPD | at 36 weeks of GA
  Composite outcome of death or BPD

CONTACTS AND LOCATIONS:
Overall Officials: Venkatakrishna Kakkilaya, MBBS, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Venkatakrishna Kakkilaya, Dallas, Texas, United States